CLINICAL TRIAL: NCT06144112
Title: A Randomized Trial Comparing the Time for Managing Intraoperative Hypofibrinogenemia Using Fibrinogen Concentrates Versus Cryoprecipitate in Liver Transplant Surgery (FIBCRYO-LT Trial)
Brief Title: Fibrinogen Concentrates Versus Cryoprecipitate in Liver Transplant Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC22195220002003
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Liver Diseases
Keywords: hypofirinogenemia; coagulopathy; fibrinogen; cryoprecipitate; liver transplantation; lyophilized factor concentrates
MeSH Terms: conditions — Liver Diseases; Hemostatic Disorders | interventions — Factor IX

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryoprecipitate (Active Comparator): If serum-fibrinogen < 100 mg/dl or CFF-MA < 15 mm in thromboelastography (TEG), cryoprecipitate is administered
  Interventions: Biological: fresh frozen plasma
- fibirnogen concentrate (Experimental): If serum-fibrinogen < 80 mg/dl or CFF-MA < 15 mm in thromboelastography (TEG), fibrinogen concentrate is administered.
  Interventions: Biological: prothrombin complex concentrate

INTERVENTIONS:
Biological: fresh frozen plasma — transfusion of fresh frozen plasma
  Arms: cryoprecipitate
Biological: prothrombin complex concentrate — prothrombin complex concentrate administration
  Arms: fibirnogen concentrate

SUMMARY:
We compared the time consumed for goal-directed management of hypofibrinogemia using two strategies during liver transplant (LT) surgery: a conventional cryoprecipitate-based strategy versus a lyophilized fibrinogen concentrate-based strategy

DETAILED DESCRIPTION:
The primary outcome is an inter-group comparison of treatment time (T-time, the duration from ordering cryoprecipitate or FC to completing its administration). The secondary measures include comparisons of perioperative bleeding, blood transfusion, coagulation profiles, reoperation, thromboembolic complications, mortality, oxygenation profiles, fibrinolysis phenotypes, and costs for bleeding management and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Liver disease undergoing Liver transplantation

Exclusion Criteria:

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
intergroup difference in the treatment time (T-time) | 1 min
  The treatment time (T-time): the duration from ordering cryoprecipitate or FC to completing its administration

SECONDARY OUTCOMES:
Red Blood Cell amount | 1 hour
  Red Blood Cell transfusion amount during surgery
FFP amount | 1 hour
  FFP transfusion amount during surgery
Platelet amount | 1 hour
  Platelet transfusion amount during surgery
r-time | 1 min
  CK r-time after PCC or FFP
CRT-MA | 1 min
  CRT-MA after PCC or FFP
CFF-MA | 1 min
  CFF-MA after PCC or FFP
Bleeding | 6 hour
  Postoperative bleeding amount
oxygenation profile | 1 hour
  PaO2/FiO2 ratio
preparation time of cryoprecipitate or FC | 1 min
  time from the start of preparation (ABO-cross matching and thawing of cryoprecipitate or unpacking FC from its storage) to the delivery to patients in the operation theater

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided